CLINICAL TRIAL: NCT03532087
Title: Explorative Trial to Identify the Impact of Denosumab on the Systemic Immunity and Local Immunologic Microenvironment in Postmenopausal Patients With HER2 Negative Breast Cancer
Brief Title: Study to Identify the Impact of Denosumab on the Immune System in Patients With HER2 Negative Breast Cancer
Acronym: PERIDENO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to new insights
Sponsor: Borstkanker Onderzoek Groep (Network)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BOOG-2017-02; 2016-005210-22 (EudraCT Number)
Record Dates: First submitted 2018-02-05; First posted 2018-05-22 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-07

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Denosumab; Chemotherapy; Immunity; Immune system; PERIDENO
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No denosumab (No Intervention): All patients undergo surgery followed by adjuvant chemotherapy. Patients in this study arm are not additionally treated with denosumab.
- Denosumab 120 mg (Experimental): All patients undergo surgery followed by adjuvant chemotherapy. Patients in this study arm are additionally treated with denosumab 120 mg every 3 weeks. First denosumab gift is before surgery, last denosumab gift is together with the last cycle of chemotherapy.
  Interventions: Drug: Denosumab 120 mg
- Denosumab 60 mg (Experimental): All patients undergo surgery followed by adjuvant chemotherapy. Patients in this study arm are additionally treated with denosumab 60 mg every 6 months. First denosumab gift is before surgery, last denosumab gift is together with the last cycle of chemotherapy.
  Interventions: Drug: Denosumab 60 mg

INTERVENTIONS:
Drug: Denosumab 120 mg — Denosumab 120 mg every 3 weeks.
  Other Names: Xgeva
  Arms: Denosumab 120 mg
Drug: Denosumab 60 mg — Denosumab 60 mg every 6 months.
  Other Names: Prolia
  Arms: Denosumab 60 mg

SUMMARY:
The aim of this prospective, randomized, multicenter, open-label, explorative phase II study is to identify the impact of (neo)adjuvant denosumab on the systemic immunity and local immunologic microenvironment in postmenopausal patients with HER2 negative non-metastatic primary breast cancer.

DETAILED DESCRIPTION:
In this study, postmenopausal patients with stage T1c + grade 3, stage II or III, HER2-negative breast cancer, which are planned to undergo surgery followed by adjuvant AC-T chemotherapy, are randomized between no denosumab, denosumab low dosing and denosumab high dosing. Denosumab administration will start one week before surgery and continue until the last chemotherapy cycle.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as 1 year without menstrual activity, previous bilateral oophorectomy, age older than 60 years or baseline FSH >20 U/l and estradiol <110 pmol/l.
* Clinical stage T1c + grade 3, stage II or III breast cancer amenable to adjuvant AC-T combination chemotherapy.
* Measurable disease (breast and/or lymph nodes).
* Histological proven HER2-negative breast cancer in the core biopsy material.
* WHO 0-2.
* Adequate bone marrow function (within 4 weeks prior to randomization): WBC≥3.0x109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l.
* Adequate liver function (within 4 weeks prior to randomization): bilirubin ≤1.5 X upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL, Alkaline Phosphatase ≤5 x UNL.
* Adequate renal function (within 4 weeks prior to randomization): the calculated creatinine clearance should be ≥50 ml/min.
* Albumin-adjusted serum calcium > 2.0 mmol/L (8.0mg/dL)
* Accessible for treatment and follow-up.
* Written informed consent.

Exclusion Criteria:

* Evidence of distant metastases (M1).
* History of breast cancer.
* Prior chemotherapy or radiation therapy.
* Previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix.
* Prior or current bisphosphonate or denosumab usage.
* Serious other diseases as recent (last 6 months) myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias.
* Current active dental problems including dental abscess or infection of the jawbone (maxilla or mandible), non-healed dental or oral surgery, a current or prior diagnosis of osteonecrosis of the jaw or planned invasive dental procedures for the course of the study.
* Known hypersensitivity reaction to any of the components of the treatment.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in intratumoral T-cell (CD4, CD8 and Treg) numbers and function between the baseline biopsy and the surgical specimen. | The change can be determined after the surgical specimen is obtained, which is around two weeks after enrolment.
  The change will be determined by use of IHC and immunofluorescent stainings.
Change in myeloid cell (M1/M2 Macrophage, MDSC, DC) numbers and function between the baseline biopsy and the surgical specimen. | The change can be determined after the surgical specimen is obtained, which is around two weeks after enrolment.
  The change will be determined by use of IHC and immunofluorescent stainings.

SECONDARY OUTCOMES:
Shift in activated T effector cell levels. | Measurements will be done in PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Shifts will be determined by comparing PBMCs (using flow cytometry) before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration.
Shift in regulatory T-cell levels. | Measurements will be done in PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Shifts will be determined by comparing PBMCs (using flow cytometry) before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration.
Change in functional response of T-cells. | Measurements will be done in PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Changes will be determined by comparing PBMCs (using stimulation tests) before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration.
Change in mature and immature myeloid cells (M1/M2 macrophage, MDSC, DC). | Measurements will be done in PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Shifts will be determined by comparing PBMCs (using flow cytometry) before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration.
Shift in myeloid cell function. | Measurements will be done in PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Shifts will be determined by comparing PBMCs (using triggering tests) before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration.
Change in stimulation capacity APCs. | Measurements will be done in PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Changes will be determined by comparing PBMCs (using restimulation tests) before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration.
Change in serum levels of RANKL and OPG. | Measurements will be done in serum from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Changes will be determined by comparing serum before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration, using ELISA.
Change in serum cytokine levels (TNF-alpha, interleukines, IFN gamma). | Measurements will be done in serum from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment.
  Changes will be determined by comparing serum before start treatment, at day of surgery before surgery and 7 days after last chemotherapy administration, using luminex.
Correlation of tumor measurements with serum measurements. | Measurements will be done in tumor material and serum from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment and tumor material from baseline and surgery.
  Measurements in tumor and serum will be correlated.
Correlation of tumor measurements with PBMCs measurements. | Measurements will be done in tumor material and PBMCs from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment and tumor material from baseline and surgery.
  Measurements in tumor and PBMCs will be correlated.
Correlation of serum measurements and PBMCs measurements. | Measurements will be done in PBMCs/serum from before start treatment, day of surgery and 7 days after last chemotherapy administration, which will be around 8 months after enrolment and tumor material from baseline and surgery.
  Measurements in serum and PBMCs will be correlated.
Toxicity according to NCI CTCAE v4.03. | Toxicity will be assessed from start treatment up to 30 days following the last dose of treatment.
  Toxicities are graded according to NCI CTCAE v4.03.
Difference in descriptive event free survival (EFS) at 3 years based on immune response. | EFS will be determined after 3 years.
  After 3 years of follow up, differences in EFS based on immune response will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Kroep, MD PhD, Principal Investigator — Leiden University Medical Center; Gerrit-Jan Liefers, MD PhD, Principal Investigator — Leiden University Medical Center; Sjoerd H van der Burg, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (8):
- Netherlands (8):
  - Ziekenhuisgroep Twente (Twenteborg ZH Almelo), Almelo
  - Gelre ziekenhuizen, Apeldoorn
  - Zuyderland Medisch Centrum (Heerlen), Heerlen
  - Spaarne Gasthuis (Hoofddorp), Hoofddorp
  - Leiden University Medical Center, Leiden
  - Fransiscus (Vlietland), Schiedam
  - VieCuri Medisch Centrum (Venlo), Venlo
  - 't Lange Land Ziekenhuis, Zoetermeer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- See also: Information PERIDENO study on BOOG website (sponsor). — https://www.boogstudycenter.nl/studie/287/perideno.html